CLINICAL TRIAL: NCT01499420
Title: A Phase 2a, Multi-center, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of a Single Intravenous Infusion of CSL112 in Patients With Stable Atherothrombotic Disease
Brief Title: A Single Ascending Dose Study Examining the Safety and Pharmacokinetic Profile of Reconstituted High Density Lipoprotein (CSL112) Administered to Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-HDL-10-70a
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Stable Atherothrombotic Disease
MeSH Terms: interventions — CSL112

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CSL112 (Experimental)
  Interventions: Biological: CSL112 (reconstituted high density lipoprotein)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSL112 (reconstituted high density lipoprotein) — Single escalating intravenous doses of CSL112
  Arms: CSL112
Biological: Placebo — Single intravenous doses of normal saline (0.9%)
  Arms: Placebo

SUMMARY:
Reconstituted high density lipoprotein used in patients with acute coronary syndrome (ACS) may reduce atherosclerotic plaque burden, thereby reducing the risk of recurrent cardiovascular events. This study is a multi-center, randomized, placebo-controlled, single ascending dose study in patients with stable atherothrombotic disease in whom the safety and pharmacokinetic profile of CSL112 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years to 80 years.
* Subjects must have documented evidence of a history of atherosclerotic coronary artery disease/surgical revascularization.
* Subjects on a stable medication regimen.
* Body weight 50 kg or greater at screening.

Exclusion Criteria:

* Moderate/severe heart failure or renal impairment.
* Uncontrolled hyperglycemia in subjects with type 1 or type 2 diabetes.
* Receipt of the combination of omeprazole and clopidogrel within 1 month of randomization.
* Subjects whose medical history, condition or medication regimen may interfere with the evaluation of the safety and tolerability of CSL112 (for example significantly altered electrocardiogram (ECG) waveform, hepatobiliary disease, malignancy, thrombocytopenia, etc.)
* Known hypersensitivity to the product components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  The frequency of study product-related adverse events
Clinically significant elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) | 14 days
  Number of subjects with clinically significant elevation of ALT or AST

SECONDARY OUTCOMES:
Pharmacokinetic profile of apolipoprotein A-I (apoA-I) | 9 days
  Plasma apoA-I concentration with and without baseline correction
Plasma apoA-I area under the curve (AUC) | 9 days
Plasma apoA-I Cmax | 9 days
Plasma apoA-I Tmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Denise D'Andrea, Study Director — CSL Limited
Locations (11):
- United States (11):
  - Study Site, Chula Vista, California
  - Study Site, Jacksonville, Florida
  - Study Site, Miami, Florida
  - Study Site, Lexington, Kentucky
  - Study Site, Madisonville, Kentucky
  - Study Site, Auburn, Maine
  - Study Site, Baltimore, Maryland
  - Study Site, Petoskey, Michigan
  - Study Site, Durham, North Carolina
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Rapid City, South Dakota

REFERENCES:
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027
- [Derived] Tricoci P, D'Andrea DM, Gurbel PA, Yao Z, Cuchel M, Winston B, Schott R, Weiss R, Blazing MA, Cannon L, Bailey A, Angiolillo DJ, Gille A, Shear CL, Wright SD, Alexander JH. Infusion of Reconstituted High-Density Lipoprotein, CSL112, in Patients With Atherosclerosis: Safety and Pharmacokinetic Results From a Phase 2a Randomized Clinical Trial. J Am Heart Assoc. 2015 Aug 25;4(8):e002171. doi: 10.1161/JAHA.115.002171. PMID 26307570